CLINICAL TRIAL: NCT01239888
Title: Phase IB Study of Efficacy and Safety of Oxytocin and Tibolone Adjuncts in Treatment Resistant Depression
Brief Title: Oxytocin and Tibolone Adjuncts in Treatment Resistant Depression - A Pilot Study
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Alfred (Other)
Collaborators: Monash University (Other)
Responsible Party: Principal Investigator, Charlotte Keating, Research Fellow, The Alfred
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MAPRC 2010CK
Record Dates: First submitted 2010-11-09; First posted 2010-11-15 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Depression; Major Depressive Disorder
Keywords: Depression; Treatment resistant depression; Oxytocin; Estrogen Modulators; HPA axis; Mental Disorders; Estrogens; Tibolone; Estrogen Receptor Modulators; Androgens; Hormones; Hormone Substitutes; Physiological Effects of Drugs; Pharmacologic Actions; Hormone Antagonists; Bone Density Conservation Agents; Estrogen Antagonists
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant; Mental Disorders | interventions — Oxytocin; tibolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Oxytocin (Active Comparator)
  Interventions: Drug: Oxytocin
- Oxytocin and Tibolone (Active Comparator)
  Interventions: Drug: Oxytocin and Tibolone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — 20 IU of intranasal oxytocin twice per day for 8 weeks, and a placebo (oral) for the 8 week trial
  Arms: Oxytocin
Drug: Oxytocin and Tibolone — 20 IU of intranasal oxytocin twice per day for 8 weeks, and 2.5mg oral tibolone for the 8 week trial
  Other Names: Livial (tibolone)
  Arms: Oxytocin and Tibolone
Drug: Placebo — 20 IU of intranasal placebo twice per day for 8 weeks, and a placebo (oral) for the 8 week trial
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether an oxytocin ad-on, or oxytocin and tibolone ad-on can induce a response to antidepressants in patients with treatment resistant depression.

DETAILED DESCRIPTION:
We are examining the efficacy and safety of oxytocin or oxytocin and tibolone with an antidepressant (SSRIs) in treatment resistant depression in a double-blind randomized clinical trial.

A secondary objective is the evaluation of neurobiological factors contributing to drug efficacy in treatment resistant depression.

ELIGIBILITY:
Inclusion Criteria:

* Women
* 18-45 years
* Current DSM-IV diagnosis of Major Depression
* Comorbid anxiety disorders secondary to depression will be included
* Past history of at least 2 failed treatment responses (including SSRIs) at the highest tolerated dose for at least 4-6 weeks
* A MADRS score >20 at randomization
* Women on a stable dose of an SSRI (sertraline, citalopram, escitalopram, paroxetine, fluoxetine or fluvoxamine) for at least 4-6 weeks.
* A negative pregnancy test at screening
* A clinically acceptable Pap smear within the past 2 years
* Must be able to use intranasal spray and swallow tablets

Patients may take up to 2 sleep medications permitted at a dose considered reasonable by the investigating team. Limited adjustments in sleep medication are acceptable. Patients will be asked to notify the researchers of any changes to their sleep medication.

Exclusion Criteria:

* Any previous history of adverse side-effects to escitalopram (or other SSRI)
* Use of oral contraceptives (or any hormonal method of contraception) for the duration of the study
* DSM-IV defined substance dependence, history of bipolar disorder, schizoaffective disorder or schizophrenia
* Significant unstable medical illness including epilepsy, diabetes or cardiac related, renal or liver disease, hormone dependent cancer or pregnancy
* A BMI<18 or > 34kg/m2
* Planning for pregnancy
* Renal disease, history of cerebrovascular disease, thrombo-embolic disorders, myocardial infarction or angina at any time before study entry or thrombo-phlebitis within the last 5 years, or any other major illness that has occurred within the last 6 months.
* An undiagnosed genital bleeding
* Moderate to severe acne or hirsutism, have used antiandrogen therapy for acne or hirsutism in the preceding 5 years, have androgenic alopecia ( will exclude women with clinically meaningful androgen excess)
* Active malignancy, or treatment for malignancy in the preceding 6 months (excluding non-melanotic skin cancer)
* Alcohol consumption in excess of 3 standard drinks per day
* Lactose intolerance
* An abnormal thyroid stimulating hormone (TSH) value at screening confirmed by a Free T4 outside the normal laboratory range (patients with an abnormal TSH, normal Free T4 and no clinical signs or symptoms of thyroid disease, with or without replacement treatment, may be admitted to the study).
* A history of allergic reactions to androgens (oral or patch)
* Chronic medications: aspirin and warfarin

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Montgomery-Asberg Depression Rating Scale (MADRS) | Assessed at different time points: 1 week, 2 weeks, 4 weeks, 8 weeks

SECONDARY OUTCOMES:
Change from baseline in Hamilton Rating Scale for Depression (HAM-D) | Assessed at different time points: 1 week, 2 weeks, 4 weeks, 8 weeks
Change from baseline in Beck Depression Inventory II (BDI-II) | Assessed at different time points: 1 week, 2 weeks, 4 weeks, 8 weeks
Change from baseline in State Trait Anxiety Inventory (STAI) | Assessed at different time points: 1 week, 2 weeks, 4 weeks, 8 weeks
Adverse Symptom Check List | baseline, week 2, week 4, week 8
Perceived stress scale | baseline, week 2, week 4, week 8
Pittsburgh sleep quality index | baseline, week 2, week 4, week 8
Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q-SF) | baseline, week 2, week 4, week 8

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Keating, PhD, Principal Investigator — Monash University and the Alfred
Locations (1):
- Monash Alfred Psychiatry Research Centre, Melbourne, Victoria, Australia